CLINICAL TRIAL: NCT04101968
Title: Multimodal Molecular Imaging and Biometric Analysis in GBA-PD and Asymptomatic GBA-mutation Carriers
Brief Title: The GBA Multimodal Study in Parkinson's Disease
Status: Recruiting | Type: Observational
Sponsor: Pacific Parkinson's Research Centre (Other)
Collaborators: University of British Columbia (Other); University of Washington (Other); Oregon Health and Science University (Other); Simon Fraser University (Other); Michael J. Fox Foundation for Parkinson's Research (Other); Silverstein Foundation (Unknown); Weston Brain Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 16451
Record Dates: First submitted 2019-09-16; First posted 2019-09-24 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Parkinson Disease; GBA Gene Mutation; Gaucher Disease
Keywords: Parkinson
MeSH Terms: conditions — Parkinson Disease; Gaucher Disease | interventions — Positron-Emission Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GBA-PD: People with Parkinson's disease who are known heterozygous carriers of pathogenic GBA gene mutations.
  Interventions: Diagnostic Test: PET scan; Diagnostic Test: neuroQWERTY
- Asymptomatic GBA: Known heterozygous carriers/obligated carriers of pathogenic GBA gene mutations.
  Interventions: Diagnostic Test: PET scan; Diagnostic Test: neuroQWERTY

INTERVENTIONS:
Diagnostic Test: PET scan — 3 PET scans to analyze the dopamine metabolism, acetylcholine and tau protein deposition in the brain.
Diagnostic Test: neuroQWERTY — Analysis of free-text typing in a computer and/or a touch-screen device.

SUMMARY:
This study plans to analyze the molecular and clinical mechanisms of the relationship between the GBA mutations and Parkinson's disease. This will be assessed through the use of advanced neuroimaging techniques called PET (positron emission tomography) to study the accumulation of the tau protein and the dysfunction of acetylcholine and dopamine in the brain of people with a mutation in the GBA gene, with and without Parkinson's disease. The ingestigators will also use a technology-based assessment to study the typing patterns as possible biomarkers of early motor dysfunctions.

DETAILED DESCRIPTION:
Study Rationale: People who have a mutation in the GBA gene have a higher risk of developing Parkinson's disease (PD) and, if they have PD, are more likely to have cognitive decline and dementia. Cognitive problems in people with PD is related to dysfunction of the brain chemical acetylcholine and likely to the accumulation of the tau protein in the brain. Another observation in previous studies is that analyzing the patterns of typing into a computer can help differentiate healthy people from people with PD.

Hypothesis: The investigators hypothesize that people with GBA-related PD will have higher acetylcholine dysfunction and tau accumulation compared with non-GBA patients, and that these changes may start in the asymptomatic phase (i.e., people with the mutation but without symptoms of PD). The investigators also believe that the investigators will be able to detect subjects with higher degree of dopamine loss just by analyzing the way they type into a computer.

Study Design: The investigators will recruit 25 subjects with a GBA mutation (10 subjects with PD and 15 asymptomatic carriers). All the participants will have a clinical evaluation and a typing session, and subsequently will undergo a brain MRI and three PET scans with a tau tracer, an acetylcholine tracer, and a dopaminergic tracer. A blood sample will also be taken for the analysis of GCase (the enzyme related to the GBA mutation).

Impact on Diagnosis/Treatment of Parkinson's Disease: The results will help understand the changes that take place in the brain of people with GBA-related Parkinson's disease, and hopefully will shed light also on the pathophysiology of non-GBA-related Parkinson's, as well as on the molecular correlates of cognitive decline, especially in its early stage. The typing data along with dopaminergic imaging will clarify the possible role of using typing patterns to identify subjects with early stage Parkinson's disease.

Next Steps for Development: The findings of this study may help identify biomarkers for cognitive decline in early Parkinson's disease, with a potential role in clinical trials. Also, if the hypothesis on the typing is confirmed, this approach may be studied in larger cohorts for early diagnosis of Parkinson's in other at-risk populations.

ELIGIBILITY:
Inclusion Criteria:

* heterozygous for a pathogenic GBA mutation (e.g., p.L444P, p.N370S) or polymorphism;
* age 18 to 80 years.

Exclusion Criteria:

* co-occurrence of other neurological disorders;
* implants that contraindicate the MRI scanning (e.g. cardiac pacemaker, ferromagnetic implants or devices);
* severe claustrophobia;
* intolerance to antiparkinsonian drug withdrawal (for GBA-PD subjects);
* ongoing treatment with cholinergic drugs

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with a known pathogenic GBA gene mutation with or without PD.
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Acetylcholinesterase activity | baseline
  11C-PMP PET
Tau protein deposition | baseline
  11C-PBB3 PET
Dopaminergic denervation | baseline
  11C-DTBZ PET
neuroQWERTY index | baseline
  Typing analysis

CONTACTS AND LOCATIONS:
Overall Officials: Michele Matarazzo, MD, Principal Investigator — Pacific Parkinson's Research Centre | University of British Columbia; A. Jon Stoessl, CM, MD, FRCPC, FCAHS, Principal Investigator — Pacific Parkinson's Research Centre | University of British Columbia
Locations (3):
- United States (2):
  - Oregon Health & Science University, Portland, Oregon
  - University of Washington, Seattle, Washington
- Pacific Parkinson's Research Centre | University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No